CLINICAL TRIAL: NCT05712980
Title: Identification of Differentially Expressed Genes in RNAseq Data of Patients With Failed Back Surgery Syndrome Treated With Different Modalities of Spinal Cord Stimulation: Looking for Biomarkers of Response and Effectiveness
Brief Title: Transcriptomic Profile of Patients Treated With Different Modalities of Spinal Cord Stimulation
Acronym: SCS-OMICS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital General Universitario de Valencia (Other)
Responsible Party: Principal Investigator, Gustavo Fabregat, Consultant of Anesthesiology and Principal Investigator, Hospital General Universitario de Valencia
Other Study IDs: SCS - OMICS
Record Dates: First submitted 2023-01-17; First posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Spinal Cord Stimulation; Failed Back Surgery Syndrome; Genetic Change
Keywords: pain; spinal cord stimulation; RNAseq; DTM; transcriptomics; omics; failed back surgery syndrome
MeSH Terms: conditions — Failed Back Surgery Syndrome; Pain | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- DTM Cohort: Patients with Failed Back Surgery Syndrome treated with Spinal Cord Stimulation with DTM programming
  Interventions: Device: Implanted pulse generator for SCS with different programming modalities
- Conventional Cohort: Patients with Failed Back Surgery Syndrome treated with Spinal Cord Stimulation with conventional programming
  Interventions: Device: Implanted pulse generator for SCS with different programming modalities

INTERVENTIONS:
Device: Implanted pulse generator for SCS with different programming modalities — Surgical technique
  Patients recruited will be scheduled for the implantation of the SCS system in two phases. The implant procedure will be performed following our standardized clinical practice under local anesthesia and moderate sedation.
  Clinical parameters
  Clinical evaluation of study subjects shall include, in addition to demographic parameters, the assessment of parameters related to pain experience, disability, quality of life, as well as other psychological variables. All these parameters will be evaluated at different times of the study.
  Sample processing
  10 ml of peripheral blood will be obtained per venopuncture at different moments, always at the same time of day and in the same anatomical location.
  Expression arrays
  After a manual removal of RNA the expression arrays and the scanning of the crystals will be carried out after hybridization

SUMMARY:
Failed Back Surgery Syndrome (FBSS) is a relatively common condition that can cause a severe disability in patients. Spinal cord stimulation (SCS) is used in those patients refractory to conventional therapies.In this project the investigators aim to identify new functional molecular basis, defined with transcriptomic profiling, differentially represented in the serum of patients suffering chronic pain caused by FBSS.

The investigators will try to Identify "omics" markers for diagnosing and monitoring the process of development and maintenance of pain as well as the evaluation of these as evolutionary disease markers or predictors of the response to SCS therapy. To carry out the project, 40 patients diagnosed with refractory FBSS and treated with an SCS system for pain management will be included. Blood samples will be obtained to analyze the transcription profiling in plasma of patients responding to different modalities of SCS therapy.

DETAILED DESCRIPTION:
Failed back surgery syndrome (FBSS) is a real challenge for the specialist because of its clinical complexity and economic importance not only in the cost of treatment but because of the high incidence of the syndrome in patients of working age and with normal life expectancy. This syndrome is a complication of lumbosacral surgery with an incidence ranging from 5-40%.

Spinal cord stimulation (SCS) has been used in the treatment of patients with FBSS for years safely and effectively . Although it was initially believed that the main mechanism of action was explained by the "Gate Control Theory" described by Wall and Melzack in 1965, it should be noted that other mechanisms beyond this could contribute to pain relief resulting from SCS. These include inhibition of neuronal excitability and hypersensitivity at the medullary level as well as changes in the release of neurotransmitters like GABA, acetylcholine, adenosine, serotonin and norepinephrine, involved in the transmission and modulation of pain. However, the molecular mechanisms underlying the therapeutic effect of SCS remain unknown.

Genetic studies are used to provide new insights into the molecular mechanisms underlying the onset and maintenance of pain. These can be driven by the hypothesis, thus evaluating the expression of default molecules, or independent of the hypothesis, exploring gene expression at the gene level at the whole genome. Microarray chips measure the expression of hundreds of genes in a given sample. Used to study a wide variety of biological systems, they have been used to evaluate extensive changes at the transcriptional level in different parts of the central or peripheral nervous system, leading to the discovery of new pain-related genes such as the Kv9.1 subunit of the potassium channel or KCNS1.

Recently, some animal model studies suggest that SCS produces extensive changes in gene expression. Tilley and collaborators found that SCS produced modulation in the expression of 5HTra, cFOS and GABAbr1 among others, with a strong correlation between the amount of current applied and the expression of GABAbr1, Na/K ATPase (negative correlation), 5HT3r and VIP (positive correlation) at the medular level and also at the level of the dorsal root ganglion. These authors focused on analyzing groups of genes that were shown altered in animal models of peripheral nerve injury. Stephens and collaborators performed an RNA seq of the spinal cord of rats with neuropathic pain secondary to the sciatic nerve ligation to which a spinal cord stimulator was implanted and found that gene expression changed after the application of SCS. They identified that the expression of some key genes in the expression of protein dense post-synaptic supporting proteins network in glutamaergic synapses is downregulated after SCS; this could destabilize this dense network, thus decreasing the effectiveness of synaptic signaling. They also found that SCS could activate nearby spinal tracts that affect neurons and gloss cells in the distal spinal segments. Vallejo and Tilley's group also performed extensive transcriptome analysis in animal models of neuropathic pain and found that SCS produces significant modulation in gene expression at the spinal cord and dorsal root ganglion level, with groups of genes and metabolic pathways similar in both tissues and which are directly or indirectly related to neural regeneration, regulation of inflammatory and immune responses and regulation of ion transport. Our group analyzed the gene expression of different markers (from cannabinoid receptors, opioid receptors and opioid peptides) using real-time polymerase chain reaction from lymphocyte RNA obtained from peripheral blood samples of patients with FBSS treated with SCS, observing a significant increase in proenkephalin (PNK) following SCS with respect to baseline levels and maintained over time.

Using the advantages of large-scale study of the genome using microarrays, we have carried out a research project in recent years with the main objective of identifying new molecular bases, defined with transcriptomic profiles, differentially expressed in the plasma of patients affected by FBSS and treated with tonic or conventional SCS. This study has been funded by Instituto de Salud Carlos III through the Project PI16/01364 (Co-funded by European Regional Development Fund/European Social Fund "A way to make Europe"/"Investing in your future"). The project was approved by the Ethical Committee for Clinical Research of the University General Hospital of Valencia. The study complied with local regulations, Good Clinical Practice guidelines, and the principles of the Declaration of Helsinki, as well as with current legislation and regulations governing protection of personal data and the rights and responsibilities regarding information and documentation in health care. Our group performed a transcriptomic analysis of the blood of patients affected of FBSS and treated with SCS (responder patients); we obtained samples before and at different times after implantation of the system in order to find differential gene expression in response to treatment and that could serve as potential biomarkers of effectiveness to therapy. We also performed transcriptomic analysis of patients in which SCS was not effective (non-responders), comparing the results with the responding patients with the intention of finding differential expression of potential biomarkers of response to SCS therapy. Finally, we compared the expression of patients diagnosed with FBSS with a group of spine-intervened patients who did not develop pain and served as a control group; we try to find differences in the gene expression between the two populations with the aim of finding possible biomarkers of disease development. We included 30 patients with SCS-treated FBSS (of whom 7 were non-responders and 23 responders) and 15 control patients. We have completed the recruitment and analysis of the samples periods and we are currently in the interpretation phase of the final results and development of the corresponding publications. Although the results are not definitive, preliminary analysis shows that there are more than 190 differentially expressed genes (p < 0.05) at baseline when comparing control patients and patients with FBSS treated with SCS. We also found more than 750 genes differentially expressed in patients implanted before and after the onset of SCS therapy.

HYPOTHESIS

The biochemical and molecular processes associated with FBSS are unknown as are the changes that occur in patients undergoing SCS. The transcriptomic analysis seem promising tools to provide insight on the mechanisms underlying chronic pain. Quantification of RNA with RT-PCR will allow to identify differential genes implicated and solid conclusions to be drawn.

Our hypothesis is based on the fact that different genetic expression must occur in clinical situations related to pain and that these alterations should be differentially modified in patients successfully treated with spinal cord stimulation.

The identification of these possible biomarkers of state or evolution of the pathology and its treatment will contribute significantly to establish more accurate therapeutic strategies and can serve as predictive biomarkers of response to treatment, guiding the selection of therapeutic targets for the development of future treatment strategies.

AIMS OF THE STUDY

Based on these hypotheses and with the hopeful results previously obtained by our group, the investigators aim to compare whether the DTM programming of the SCS system produces a different expression-level effect than conventional programming with the intention of seeking biomarkers of response and evolution to this programming modality.

The investigators also aim to study whether these differences could be in relation to significantly different clinical outcomes and correlate with the intensity of the effect of the different modalities.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients affected by FBSS, defined as "surgical end stage after one or several interventions on the lumbar neuroaxis indicated to relief lower back pain, root pain or the combination of both, without effect"
* Age between 18 and 65 years
* Severe pain measured on a numerical rating scale (NRS > 6/10), more than six months of evolution
* Refractory pain despite having carried out pharmacological treatment according to WHO's stratified approach; physical/rehabilitation therapy and/or interventional procedures (e.g. epidural steroid injections, radiofrequency, epiduroscopy/adhesiolysis)

Exclusion Criteria:

* Patients with severe associated comorbidities (e.g. severe high blood pressure, diabetes mellitus, peripheral vasculopathy, severe heart disease, etc...) that may in themselves cause pain or aggravate the existence of previous pain.
* Extensive osteosynthesis encompassing the thoraco-lumbar region where the tips of the electrodes are routinely positioned.
* Abnormal pain behavior, unresolved psychiatric illness, unresolved issues of secondary gain or inappropriate medication use
* Patients not consenting or refusing to participate will be excluded
* Negative evaluation of the psychologist previous to the implant

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients affected by FBSS fullfilling all the inclusion and none of the exclusion criteria will be included.
  Following our usual protocol, all patients will attend a session with our psychologist to consider the adequacy of the treatment to be used and to determine the effect of psychosocial issues on their pain complaints. A negative evaluation will be considered a key exclusion criterion. Patients will be instructed to keep their medication dosage stable throughout the study.
  All the subjects of study will be implanted with the same device from Medtronic. The device will be programmed with two different strategies, the conventional one and the Differential Targeted Multiplexed (DTM) programming.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Transcriptomic profile change in DTM responders | T0: Before IPG; T1: 15 days after IPG and T2 2 months after IPG
  Identify the transcriptomic signature of responding patients undergoing DTM programming of the SCS system and analyze potential changes over time

SECONDARY OUTCOMES:
DTM vs Conventional signatures | T0: Before IPG; T1: 15 days after IPG and T2 2 months after IPG
  Compare whether the DTM programming of the SCS system produces a different expression-level effect than conventional programming
Transcriptomic Profile vs Clinical Outcomes | T0: Before IPG; T1: 15 days after IPG and T2 2 months after IPG
  Analyze potential correlations between the transcriptomic profiles measured wiht RNAseq techniques with clinical measurements (Intensity of pain measured with Numeric Rating Scale and level of disability measured with Oswestry Scale
Intensity of pain | T0: Before IPG; T1: 15 days after IPG and T2 2 months after IPG
  Measure the intensity of pain with a Numeric Rating Scale (NRS) in different moments before and after the treatment with SCS
QOL | T0: Before IPG; T1: 15 days after IPG and T2 2 months after IPG
  Measure the quality of life of patients with FBSS who undergo treatment with a spinal cord stimulation system with the SF12 questionnaire in different moments before and after the treatment with SCS
Level of disability | T0: Before IPG; T1: 15 days after IPG and T2 2 months after IPG
  Measure the Level of disability of patients with FBSS who undergo treatment with a spinal cord stimulation system with the Oswestry Score in different moments before and after the treatment with SCS

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Fabregat, MD, PhD, Principal Investigator — Consultant of Anesthesiology and Pain Medicine Department
Locations (1):
- Consorcio Hospital General Universitario, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gybels J, Erdine S, Maeyaert J, Meyerson B, Winkelmuller W, Augustinsson L, Bonezzi C, Brasseur L, DeJongste M, Kupers R, Marchettini P, Muller-Schwefe G, Nitescu P, Plaghki L, Reig E, Spincemaille G, Thomson S, Tronnier V, Van Buyten JP. Neuromodulation of pain. A consensus statement prepared in Brussels 16-18 January 1998 by the following task force of the European Federation of IASP Chapters (EFIC). Eur J Pain. 1998;2(3):203-9. doi: 10.1016/s1090-3801(98)90016-7. No abstract available. PMID 15102380
- [Background] Gonzalez Viejo MA, Condon Huerta MJ. [Disability from low back pain in Spain]. Med Clin (Barc). 2000 Apr 8;114(13):491-2. doi: 10.1016/s0025-7753(00)71342-x. Spanish. PMID 10846653
- [Background] Turner JA, Loeser JD, Deyo RA, Sanders SB. Spinal cord stimulation for patients with failed back surgery syndrome or complex regional pain syndrome: a systematic review of effectiveness and complications. Pain. 2004 Mar;108(1-2):137-47. doi: 10.1016/j.pain.2003.12.016. PMID 15109517
- [Background] Van Buyten JP. Neurostimulation for chronic neuropathic back pain in failed back surgery syndrome. J Pain Symptom Manage. 2006 Apr;31(4 Suppl):S25-9. doi: 10.1016/j.jpainsymman.2005.12.012. PMID 16647592
- [Background] Inoue S, Kamiya M, Nishihara M, Arai YP, Ikemoto T, Ushida T. Prevalence, characteristics, and burden of failed back surgery syndrome: the influence of various residual symptoms on patient satisfaction and quality of life as assessed by a nationwide Internet survey in Japan. J Pain Res. 2017 Apr 6;10:811-823. doi: 10.2147/JPR.S129295. eCollection 2017. PMID 28435318
- [Background] Taylor RS, Taylor RJ. The economic impact of failed back surgery syndrome. Br J Pain. 2012 Nov;6(4):174-81. doi: 10.1177/2049463712470887. PMID 26516490
- [Background] Chan CW, Peng P. Failed back surgery syndrome. Pain Med. 2011 Apr;12(4):577-606. doi: 10.1111/j.1526-4637.2011.01089.x. Epub 2011 Apr 4. PMID 21463472
- [Background] North RB, Wetzel FT. Spinal cord stimulation for chronic pain of spinal origin: a valuable long-term solution. Spine (Phila Pa 1976). 2002 Nov 15;27(22):2584-91; discussion 2592. doi: 10.1097/00007632-200211150-00035. PMID 12435997
- [Background] Kumar K, Taylor RS, Jacques L, Eldabe S, Meglio M, Molet J, Thomson S, O'Callaghan J, Eisenberg E, Milbouw G, Buchser E, Fortini G, Richardson J, North RB. Spinal cord stimulation versus conventional medical management for neuropathic pain: a multicentre randomised controlled trial in patients with failed back surgery syndrome. Pain. 2007 Nov;132(1-2):179-88. doi: 10.1016/j.pain.2007.07.028. Epub 2007 Sep 12. PMID 17845835
- [Background] Melzack R, Wall PD. Pain mechanisms: a new theory. Science. 1965 Nov 19;150(3699):971-9. doi: 10.1126/science.150.3699.971. No abstract available. PMID 5320816
- [Background] Zhang TC, Janik JJ, Grill WM. Mechanisms and models of spinal cord stimulation for the treatment of neuropathic pain. Brain Res. 2014 Jun 20;1569:19-31. doi: 10.1016/j.brainres.2014.04.039. Epub 2014 May 4. PMID 24802658
- [Background] Zhang TC, Janik JJ, Peters RV, Chen G, Ji RR, Grill WM. Spinal sensory projection neuron responses to spinal cord stimulation are mediated by circuits beyond gate control. J Neurophysiol. 2015 Jul;114(1):284-300. doi: 10.1152/jn.00147.2015. Epub 2015 May 13. PMID 25972582
- [Background] Linderoth B, Foreman RD. Conventional and Novel Spinal Stimulation Algorithms: Hypothetical Mechanisms of Action and Comments on Outcomes. Neuromodulation. 2017 Aug;20(6):525-533. doi: 10.1111/ner.12624. Epub 2017 May 31. PMID 28568898
- [Background] Guan Y, Wacnik PW, Yang F, Carteret AF, Chung CY, Meyer RA, Raja SN. Spinal cord stimulation-induced analgesia: electrical stimulation of dorsal column and dorsal roots attenuates dorsal horn neuronal excitability in neuropathic rats. Anesthesiology. 2010 Dec;113(6):1392-405. doi: 10.1097/ALN.0b013e3181fcd95c. PMID 21068658
- [Background] Shechter R, Yang F, Xu Q, Cheong YK, He SQ, Sdrulla A, Carteret AF, Wacnik PW, Dong X, Meyer RA, Raja SN, Guan Y. Conventional and kilohertz-frequency spinal cord stimulation produces intensity- and frequency-dependent inhibition of mechanical hypersensitivity in a rat model of neuropathic pain. Anesthesiology. 2013 Aug;119(2):422-32. doi: 10.1097/ALN.0b013e31829bd9e2. PMID 23880991
- [Background] Yang F, Xu Q, Cheong YK, Shechter R, Sdrulla A, He SQ, Tiwari V, Dong X, Wacnik PW, Meyer R, Raja SN, Guan Y. Comparison of intensity-dependent inhibition of spinal wide-dynamic range neurons by dorsal column and peripheral nerve stimulation in a rat model of neuropathic pain. Eur J Pain. 2014 Aug;18(7):978-88. doi: 10.1002/j.1532-2149.2013.00443.x. Epub 2014 Jan 6. PMID 24390782
- [Background] Stiller CO, Cui JG, O'Connor WT, Brodin E, Meyerson BA, Linderoth B. Release of gamma-aminobutyric acid in the dorsal horn and suppression of tactile allodynia by spinal cord stimulation in mononeuropathic rats. Neurosurgery. 1996 Aug;39(2):367-74; discussion 374-5. doi: 10.1097/00006123-199608000-00026. PMID 8832675
- [Background] Cui JG, O'Connor WT, Ungerstedt U, Linderoth B, Meyerson BA. Spinal cord stimulation attenuates augmented dorsal horn release of excitatory amino acids in mononeuropathy via a GABAergic mechanism. Pain. 1997 Oct;73(1):87-95. doi: 10.1016/s0304-3959(97)00077-8. PMID 9414060
- [Background] Schechtmann G, Song Z, Ultenius C, Meyerson BA, Linderoth B. Cholinergic mechanisms involved in the pain relieving effect of spinal cord stimulation in a model of neuropathy. Pain. 2008 Sep 30;139(1):136-145. doi: 10.1016/j.pain.2008.03.023. Epub 2008 May 9. PMID 18472215
- [Background] Cui JG, Meyerson BA, Sollevi A, Linderoth B. Effect of spinal cord stimulation on tactile hypersensitivity in mononeuropathic rats is potentiated by simultaneous GABA(B) and adenosine receptor activation. Neurosci Lett. 1998 May 15;247(2-3):183-6. doi: 10.1016/s0304-3940(98)00324-3. PMID 9655623
- [Background] Linderoth B, Gazelius B, Franck J, Brodin E. Dorsal column stimulation induces release of serotonin and substance P in the cat dorsal horn. Neurosurgery. 1992 Aug;31(2):289-96; discussion 296-7. doi: 10.1227/00006123-199208000-00014. PMID 1381066
- [Background] LaCroix-Fralish ML, Austin JS, Zheng FY, Levitin DJ, Mogil JS. Patterns of pain: meta-analysis of microarray studies of pain. Pain. 2011 Aug;152(8):1888-1898. doi: 10.1016/j.pain.2011.04.014. Epub 2011 May 10. PMID 21561713
- [Background] Tsantoulas C, Zhu L, Shaifta Y, Grist J, Ward JP, Raouf R, Michael GJ, McMahon SB. Sensory neuron downregulation of the Kv9.1 potassium channel subunit mediates neuropathic pain following nerve injury. J Neurosci. 2012 Nov 28;32(48):17502-13. doi: 10.1523/JNEUROSCI.3561-12.2012. PMID 23197740
- [Background] Costigan M, Belfer I, Griffin RS, Dai F, Barrett LB, Coppola G, Wu T, Kiselycznyk C, Poddar M, Lu Y, Diatchenko L, Smith S, Cobos EJ, Zaykin D, Allchorne A, Gershon E, Livneh J, Shen PH, Nikolajsen L, Karppinen J, Mannikko M, Kelempisioti A, Goldman D, Maixner W, Geschwind DH, Max MB, Seltzer Z, Woolf CJ. Multiple chronic pain states are associated with a common amino acid-changing allele in KCNS1. Brain. 2010 Sep;133(9):2519-27. doi: 10.1093/brain/awq195. Epub 2010 Aug 18. PMID 20724292
- [Background] Tilley DM, Cedeno DL, Kelley CA, Benyamin R, Vallejo R. Spinal Cord Stimulation Modulates Gene Expression in the Spinal Cord of an Animal Model of Peripheral Nerve Injury. Reg Anesth Pain Med. 2016 Nov/Dec;41(6):750-756. doi: 10.1097/AAP.0000000000000452. PMID 27512935
- [Background] Tilley DM, Cedeno DL, Kelley CA, DeMaegd M, Benyamin R, Vallejo R. Changes in Dorsal Root Ganglion Gene Expression in Response to Spinal Cord Stimulation. Reg Anesth Pain Med. 2017 Mar/Apr;42(2):246-251. doi: 10.1097/AAP.0000000000000550. PMID 28079752
- [Background] Vallejo R, Tilley DM, Williams J, Labak S, Aliaga L, Benyamin RM. Pulsed radiofrequency modulates pain regulatory gene expression along the nociceptive pathway. Pain Physician. 2013 Sep-Oct;16(5):E601-13. PMID 24077210
- [Background] Vallejo R, Tilley DM, Cedeno DL, Kelley CA, DeMaegd M, Benyamin R. Genomics of the Effect of Spinal Cord Stimulation on an Animal Model of Neuropathic Pain. Neuromodulation. 2016 Aug;19(6):576-86. doi: 10.1111/ner.12465. Epub 2016 Jul 8. PMID 27391866
- [Background] De Andres J, Navarrete-Rueda F, Fabregat G, Garcia-Gutierrez MS, Monsalve-Dolz V, Harutyunyan A, Minguez-Marti A, Rodriguez-Lopez R, Manzanares J. Differences in Gene Expression of Endogenous Opioid Peptide Precursor, Cannabinoid 1 and 2 Receptors and Interleukin Beta in Peripheral Blood Mononuclear Cells of Patients With Refractory Failed Back Surgery Syndrome Treated With Spinal Cord Stimulation: Markers of Therapeutic Outcomes? Neuromodulation. 2021 Jan;24(1):49-60. doi: 10.1111/ner.13111. Epub 2020 Feb 6. PMID 32027775
- [Background] Sakai A, Suzuki H. Emerging roles of microRNAs in chronic pain. Neurochem Int. 2014 Nov;77:58-67. doi: 10.1016/j.neuint.2014.05.010. Epub 2014 Jun 3. PMID 24905749
- [Background] Monsalve V, de Andres JA, Valia JC. Application of a psychological decision algorithm for the selection of patients susceptible to implantation of neuromodulation systems for the treatment of chronic pain. A proposal. Neuromodulation. 2000 Oct;3(4):191-200. doi: 10.1046/j.1525-1403.2000.00191.x. PMID 22151524
- [Background] De Andres J, Monsalve-Dolz V, Fabregat-Cid G, Villanueva-Perez V, Harutyunyan A, Asensio-Samper JM, Sanchis-Lopez N. Prospective, Randomized Blind Effect-on-Outcome Study of Conventional vs High-Frequency Spinal Cord Stimulation in Patients with Pain and Disability Due to Failed Back Surgery Syndrome. Pain Med. 2017 Dec 1;18(12):2401-2421. doi: 10.1093/pm/pnx241. PMID 29126228